CLINICAL TRIAL: NCT00000368
Title: Treatment of Panic Disorder: Long Term Strategies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Natalia A. Skritskaya, PhD, Co-investigator, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH045964 (NIH); R01MH045964 (NIH); R01MH045965 (NIH); R01MH045966 (NIH); R01MH045963 (NIH); DSIR AT-CT
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Panic Disorder; Agoraphobia
Keywords: Adult; Cognitive Behavioral Therapy; Pharmacotherapy; Long term treatment; Remission and relapse; Male; Panic Disorder; Paroxetine; Serotonin Uptake Inhibitors; Panic Disorder -- *therapy; Panic Disorder -- drug therapy; Paroxetine -- *therapeutic use; Serotonin Uptake Inhibitors -- *therapeutic use
MeSH Terms: conditions — Panic Disorder; Agoraphobia; Recurrence | interventions — Cognitive Behavioral Therapy; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Cognitive behavior therapy
Drug: Paroxetine or other medication - algorithm used

SUMMARY:
Cognitive behavior therapy (CBT) with or without medication has been used in the treatment of panic disorder (PD). The purpose of this study is 1) to determine whether nine months of maintenance cognitive-behavior therapy (CBT) significantly improves the likelihood of sustained improvement; and 2) to determine the acute acceptability and efficacy of medication therapy or continued CBT alone among patients who fail to respond sufficiently to an initial course of CBT alone.

It has been found that patients with PD respond as well to CBT or medication alone as they do to a combination of the two. Since the combined treatments are expensive and CBT is associated with less risk of medical toxicity compared to medications, CBT alone will be used first.

All patients will first receive CBT alone. If the patient responds to this therapy, the patient will be assigned randomly (like tossing a coin) to 1 of 2 groups. One group will continue to receive CBT (maintenance therapy) for 9 months. The other group of responders will not receive any further therapy. If a patient does not respond to CBT alone, he/she will be assigned randomly to 1 of 2 different groups. One group will receive paroxetine; the other will continue to receive CBT for a longer period. The response to treatment will be evaluated to see which regimen works best to treat PD. The study will last approximately 3 years.

An individual may be eligible for this study if he/she has panic disorder with no more than mild agoraphobia (fear of being in public places) and is at least 18 years old.

DETAILED DESCRIPTION:
To determine if maintenance CBT produces a more sustained improvement among patients with panic disorder (PD) who respond to an initial course of cognitive behavior therapy (CBT) alone. For those who do not respond sufficiently to CBT alone, to determine if the addition of pharmacotherapy is acceptable and if this improves response among those inadequate responders to CBT alone.

This multicenter study builds upon the findings of a prior study comparing imipramine, placebo, CBT, and their combination in the treatment of PD patients with no more than mild agoraphobia. That study found response rates were as high with CBT or imipramine alone as with their combination. Given the added cost of combined treatments, it therefore seems reasonable to begin with monotherapy. Further, following general principles of medical practice, it would be reasonable to initiate treatment with the less invasive cognitive behavioral intervention. It is then important to learn what should be done following initial treatment.

All patients initially receive CBT alone. Patients are then randomized into 1 of 2 post-acute studies, depending on response status. Responders are randomized to a maintenance study comparing no maintenance with 9 months of continued CBT. Nonresponders are randomized to a study comparing paroxetine with continued CBT. The following outcomes will be examined: the necessity of maintenance therapy in maintaining response; the ability of adjunct pharmacotherapy to improve the response of patients who did not respond to CBT alone; possible predictors of response and relapse; and possible mediators of response.

ELIGIBILITY:
Inclusion Criteria:

- primary diagnosis of Panic disorder with or without Agoraphobia (all levels of agoraphobia are included).

Exclusion Criteria:

* current substance abuse or dependence,
* current active suicidal potential;
* any history of psychosis, bipolar disorder (I or II) or cyclothymia;
* pending application or existing medical disability claim;
* significant cognitive impairment,
* current uncontrolled general medical illness requiring intervention,
* psychotherapy directed at anxiety or panic which will not be discontinued by the first treatment visit, and daily use of 2mg of Xanax or equivalent.

Exclusion criteria for paroxetine study:

* hypersensitivity to Selective Serotonin Reuptake Inhibitors (SSRI),
* pregnancy, lactation, or planned pregnancy during the course of the study,
* contemporaneous medication that may interfere or interact with paroxetine,
* prior treatment with therapeutic doses of paroxetine (40mg/d for 1 mo),
* concurrent treatment with antidepressants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 1999-02; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Panic Disorder Severity Scale | At baseline and major assessment points plus monthly.
  This is a 7-item scale providing ratings of core features of panic disorder and the degree of work and social impairment/interference due to the disorder.
Clinical Global Impressions | Monthly, including all nonpretreatment major assessments.
  Commonly used global rating of improvement.

SECONDARY OUTCOMES:
Albany Panic and Phobia Questionnaire | All major assessment points.
  This is a 27-item scale consisting of three subscales that assess fear of agoraphobic situations, social situations, and situations and activities that produce bodily sensations commonly feared by individuals with panic disorder.
Anxiety Sensitivity Index | All major assessments and treatment visits.
  This is a 16-item scale that assesses person's tendency to regard physiologic arousal as harmful.
Subjective Symptoms Scale | All major assessment points
  This is an individual's rating of the extent to which anxiety symptoms interfere with five areas of daily functioning: work, home management, private leisure, social leisure, and family relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine H. Shear, MD, Study Chair — University of Pittsburgh; David H Barlow, PhD, Principal Investigator — Boston University Department of Psychology; Jack Gorman, MD, Principal Investigator — Columbia University School of Medicine; Scott Woods, MD, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Yale University, Department of Psychiatry, Anxiety Disorders Research Clinic, New Haven, Connecticut
  - Boston University, Department of Psychology, Center for Anxiety and Related Disorders, Boston, Massachusetts
  - Hillside Hospital Phobia Clinic, New York, New York
  - University of Pittsburgh, Department of Psychiatry, Panic, Anxiety and Traumatic Grief Program, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Barlow DH, Gorman JM, Shear MK, Woods SW. Cognitive-behavioral therapy, imipramine, or their combination for panic disorder: A randomized controlled trial. JAMA. 2000 May 17;283(19):2529-36. doi: 10.1001/jama.283.19.2529. PMID 10815116
- [Background] Shear MK, Brown TA, Barlow DH, Money R, Sholomskas DE, Woods SW, Gorman JM, Papp LA. Multicenter collaborative panic disorder severity scale. Am J Psychiatry. 1997 Nov;154(11):1571-5. doi: 10.1176/ajp.154.11.1571. PMID 9356566
- [Background] Gorman JM. A 28-year-old woman with panic disorder. JAMA. 2001 Jul 25;286(4):450-7. doi: 10.1001/jama.286.4.450. No abstract available. PMID 11466124
- [Background] Grilo CM, Money R, Barlow DH, Goddard AW, Gorman JM, Hofmann SG, Papp LA, Shear MK, Woods SW. Pretreatment patient factors predicting attrition from a multicenter randomized controlled treatment study for panic disorder. Compr Psychiatry. 1998 Nov-Dec;39(6):323-32. doi: 10.1016/s0010-440x(98)90043-8. PMID 9829138
- [Background] Huppert JD, Bufka LF, Barlow DH, Gorman JM, Shear MK, Woods SW. Therapists, therapist variables, and cognitive-behavioral therapy outcome in a multicenter trial for panic disorder. J Consult Clin Psychol. 2001 Oct;69(5):747-55. doi: 10.1037//0022-006x.69.5.747. PMID 11680551
- [Background] Hofmann SG, Barlow DH, Papp LA, Detweiler MF, Ray SE, Shear MK, Woods SW, Gorman JM. Pretreatment attrition in a comparative treatment outcome study on panic disorder. Am J Psychiatry. 1998 Jan;155(1):43-7. doi: 10.1176/ajp.155.1.43. PMID 9433337
- [Derived] Payne LA, White KS, Gallagher MW, Woods SW, Shear MK, Gorman JM, Farchione TJ, Barlow DH. SECOND-STAGE TREATMENTS FOR RELATIVE NONRESPONDERS TO COGNITIVE BEHAVIORAL THERAPY (CBT) FOR PANIC DISORDER WITH OR WITHOUT AGORAPHOBIA-CONTINUED CBT VERSUS SSRI: A RANDOMIZED CONTROLLED TRIAL. Depress Anxiety. 2016 May;33(5):392-9. doi: 10.1002/da.22457. Epub 2015 Dec 10. PMID 26663632
- See also: Center for Anxiety and Related Disorders [Boston Study Site] — http://www.bu.edu/anxiety/
- See also: Yale Anxiety Disorders Research Clinic [New Haven Study site] — http://info.med.yale.edu/yfp/new/anxiety.html